CLINICAL TRIAL: NCT06682650
Title: PB-iCRC: Multi-site Practice-Based Implementation of a ColoRectal Cancer Screening Intervention
Brief Title: Implementation of a ColoRectal Cancer Screening Tool in US Primary Care Practices - Usual Quality Improvement (10 Clinics) vs Normalization Process Theory-Participatory Learning in Action (10 Clinics)
Acronym: (PB-iCRC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); DARTNet Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00150145; R01CA289772 (NIH)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Carcinoma
Keywords: colorectal carcinoma; implementation science; cancer prevention; cancer screening; normalization process theory; participatory health research; cluster randomized trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective parallel cluster randomized trial, in which clinics are units of randomization (10 in active intervention, 10 in active comparator), and nested within clinics individual patient enrollees (whose CRC screening outcomes are Aim 1 outcomes of the study), and implementation team participants (whose survey and qualitative interview data are Aim 2 outcomes of the study).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual QI (Active Comparator): I-teams in each Usual QI clinic will be provided a pre-set protocol to implement the I2 tool into routine clinic CRC screening workflow (which they will define via a provided checklist). The protocol instructs the clinic to provide access to I2 zero to two weeks before a clinic visit, review the patient's I2 screening intentions with the patient in the clinic visit, at which time staff will order and schedule CRC screening in the visit. I2 may be completed on-line or via a paper form. I-teams will meet monthly to make progress on their implementation of I2, and complete a report/meet a study staff member monthly (separately) to report on their meetings and progress but will not receive coaching or skill training.
  Interventions: Behavioral: Usual Quality Improvement
- NPT-PLA (Experimental): Clinics randomized to NPT-PLA will also define their CRC screening workflow via a checklist and preset I2 implementation protocol but will be trained initially then receive monthly support to facilitate a "Participatory Learning in Action" (PLA) session. NPT-PLA i-teams will identify barriers and supports to I2 implementation, and use Normalization Process Theory (NPT) constructs to guide identification, selection and ordering of action steps to progress implementation e.g. "(before taking the step) does everyone understand the step to be taken, does everyone who needs to act 'buy in', (during implementation of the step) is everyone who needs to act actually taking action to complete the step, (after the step is taken) did taking the step have the intended impact, if not what happened?" . NPT-PLA I-teams can adapt the I2 implementation protocol to fit their context, including when and how patients are presented with I2, to maximize I2 implementation and CRC screening completion.
  Interventions: Behavioral: NPT-PLA

INTERVENTIONS:
Behavioral: NPT-PLA — NPT-PLA was developed and initially tested in 5 European countries in the EU-funded RESTORE study. PLA "Participatory Learning in Action" is a set of participatory research techniques in which participants use democratic processes to identify key actions needed to achieve a specific goal e.g. implementation of a tested decision making tool such as I2; and prioritize which of these need to be acted upon first and subsequently (in which order). Normalization Process Theory (NPT) is combined with PLA to help implementation teams using PLA to assess organization capacity and readiness to enact the selected action steps vis-a-vis NPT constructs, iteratively. These are coherence "does everyone understand what needs to be done?"; Cognitive participation "Does everyone who needs to act 'buy in' to take action"; collective action "Is everyone who needs to act taking steps to make the change?'; and reflexive monitoring "After the step has been taken, has it had the desired impact on the goal?"
  Arms: NPT-PLA
Behavioral: Usual Quality Improvement — Usual quality improvement includes principles of continuous quality improvement, such as Plan-Do-Study-Act cycles, to implement a specific goal. In this study, 'usual QI' methods already in use in 'active comparator' arm will be documented during the baseline assessment of clinical workflows in clinics assigned to that arm; and will be provided with a 'preset protocol' to implement the study shared decision-making tool (I2). Processes that implementation teams in these clinics use to achieve implementation will be documented.
  Arms: Usual QI

SUMMARY:
Although implementation intentions (I2)-based tools enhance colorectal cancer (CRC) screening uptake, prior studies have not tested their implementation into routine primary care delivery. In this study, investigators will conduct a cluster-randomized trial in 20 US primary care clinics. Specific aims for the project will be: 1) to test whether a Normalization Process Theory-informed Participatory Learning in Action (NPT-PLA intervention) implementation of a proven implementation Intentions-based colorectal cancer screening tool ("I2") improves screening uptake (i.e. screening order and completion) within 6 months of patient enrollment versus usual quality improvement (control) implementation; and 2) to evaluate the facilitators and barriers of each implementation arm using the 2022 expanded Normalization Process Theory (NPT) framework. Multi-disciplinary clinic 'implementation teams' that include clinic staff and patients whose preferred language is Spanish will meet monthly during the first 6 months of clinic participation and aim to integrate into routine primary care the "I2" CRC screening tool, using the NPT-PLA intervention or control approach. The I2 tool addresses the "when," "where" and "how" details of stool sample or colonoscopy screening. The I2 tool will be delivered via an on-line survey or (if patients prefer) by paper form customized for use in English or Spanish. At least 100 patients in each clinic will be enrolled in the first 6 months of clinic participation (2000 in total). All patients eligible for CRC screening will be offered the I2 tool. Their choices will be communicated automatically to clinics for order entry. Primary (Aim 1) outcomes will be CRC screening orders placed (by clinic staff); completion of the I2 tool and CRC screening completion (by patients) over 6 months of patient follow-up. For Aim 2, surveys based on the NPT domains (the "NOMAD") will be used to assess staff comprehension of their role in implementing the I2-based CRC screening tool, its salience, their buy-in, feasibility of altering workflows, and the potential impact of using the tool in their setting. Investigators will conduct summative qualitative focus group discussions in all participating clinics after 6 months of clinic participation. The study will provide important information on barriers and facilitators of embedding NPT-PLA interventions in "real-world" primary care clinical settings.

DETAILED DESCRIPTION:
The study is a Type 3 Hybrid cluster-randomized trial to be conducted in 20 practices that are members of the DARTNet Institute/American Academy of Family Physicians National Research Network. Investigators will use this approach because the implementation intervention they are testing is delivered at the clinic level; and because they have already tested the I2- tool that they are implementing and found it is effective. Clinics will be randomly assigned to 1 of the 2 study arms (NPT-PLA or usual QI 'control'), so that neither clinic staff nor DARTNet/AAFP NRNstudy staff know in advance the arm to which a clinic will be assigned. Clinics will each participate for one year. Clinics will enter the study over the first 3 years of the study in a rolling fashion, starting in the 4th quarter of year 1 (2 clinics randomized 1:1 every 3 months thereafter until all have been enrolled), with a maximum of 8 clinics simultaneously participating at any one time.

Individual patients needing CRC screening will be enrolled in the first 6 months ("active intervention" period) of a clinic's participation and followed for 6 months after they are provided access to the I2 screening tool (between inception and 6 months during the period of clinic participation), to monitor if they used the tool, and if CRC screening was ordered and completed.

During the active intervention period (first 6 months of participation), all clinics in both arms will form clinic-based 'implementation teams' that will meet monthly to plan how they will implement the I2 tool. On entry to the study, each clinic will work with DARTNet staff in both arms of the study to produce a workflow map that describes how they currently conduct CRC screening. Control clinics will be provided a prespecified workflow (the "pilot protocol") that follows the approach that the investators developed in our 2019-22 pilot study; and asked to integrate the I2 tool into their existing clinic workflow. NPT-PLA clinics will also be given the pilot protocol, but they will also use a survey-based assessments of their clinic's capacity to implement the I2 tool using the NPT based NOMAD tool. Control clinics will also complete this, but will not use the results to guide 'usual QI' processes in their clinic. Thereafter, intervention teams will meet monthly to adapt the pilot protocol using NPT-PLA methods and use their adapted approach to implement the I2 tool in their clinical context. Finally, the investigators will use NPT (2022) informed qualitative interviews at the end of the active intervention in all participating clinics to conduct a summative evaluation of the implementation process.

Study arms and interventions are further described in that section of this Record

Twenty clinics will be randomly assigned 1:1 to treatment group (NPT-PLA -10 clinics) or 'usual QI' (10 clinics) at the time of the clinic's study entry (which will take place during the first 4 years of the study), based on random numbers generated by study biostatisticians and delivered to DARNet/AAFP NRN study staff responsible for recruitment and enrollment. Randomization will be determined using covariate-adaptive randomization, a statistical technique that will help balance participants' characteristics other than the different interventions they experience. Study biostatisticians who analyze the study data will not be told which clinics are in which treatment group. Each clinic will participate for a total of 12 months. Clinics will be recruited via email and a one-page description of the project.

Clinic 'implementation team' members Clinic staff and patients in both treatment groups will participate in clinic-based "implementation teams" ("iteams").

Investigators will recruit clinic staff members (front desk staff, nursing assistants, LPNs, RNs, physicians and representative patients) to participate in each clinic's 'implementation team'. Patients will be identified by clinic managers, and invited via email/patient portal to participate in the clinic's implementation team. NOTE: since patients who participate in implementation teams will differ from other patients of the clinic in terms of their awareness of and motivation to complete I2, investigators will not include their CRC screening related outcomes in our analytic data set; however, they will be demographically similar to patients of the clinic who are eligible for CRC screening and will have access to the I2 tool for their own use. . All staff and patients participating in these implementation teams will provide written informed consent.

Patients whose CRC outcomes are monitored (within assigned clinic) To address Aim 1 outcomes, CRC screening outcomes will be monitored for clinic patients eligible for CRC screening. Please see the Eligibility section for inclusion/exclusion criteria for these patients. Each clinic will receive a list of eligible patients that is created from that clinic's EMR. This will be extracted by our contractor DARTNet. Once a list of eligible patients has been created for each clinic on the basis of this data, the list will be provided by DARTNet to that clinic. This list will indicate which patients age into or out of the eligible age range during the first 6 months of clinic participation, so that those who have not completed I2 or have ordered/completed CRC screens can be presented with the I2 tool, appropriately. Those patients not excluded will be considered "enrolled". Each clinic will enroll at least 100 patients; however, investigators will aim to enroll all who are eligible to be screened. Each patient will be followed for 6 months after their initial invitation to complete I2.

Delivery of Intervention Please see "Arms and Interventions" Section for a description of the study arms and associated intervention.

After assignment to 1 of the 2 study arms and collection of baseline survey data, clinics in each arm will start to meet to discuss how to implement the I2 tool. Prior to the initial meeting, Team Leads at each site in both arms (the Practice Manager, Head Nurse or Lead Physician) will complete a checklist to identify: how CRC screening eligible patients are identified and when; how and when screening options are presented and decided upon; if and how patient navigation occurs after screening recommendations are made for each type of screening test; how barriers and/or facilitators at different stages in clinical workflows alter clinician orders and/or patient completion of CRC screening; and what QI methods the clinic uses to monitor and optimize CRC screening, including for patients whose preferred language is Spanish. DARTNet/ AAFP NRN Study staff will use this information to create a 'workflow map' describing how the clinic carries out CRC screening for it's patients. Each team will start their discussions based on a prescribed protocol to implement I2 in their clinic workflow.

NPT-PLA (active intervention) clinics Team Leads will be trained to facilitate PLA meetings,informed by a summary of their team's NOMAD scores, which score is derived from 23 Likert-style questions (range 0-10 indicating agreement to the statement) that correspond to NPT core constructs. Usual QI (control) clinic Team Leads will use their usual 'quality improvement' methods to follow the 'pilot protocol' as closely as possible .

Teams in both arms of the trial will meet monthly for 6 months, following their respective approaches (NPT-PLA or usual QI) to increase I2 tool use by patients and CRC screening overall. In the 6th month, teams in both arms will take the NOMAD survey. In the 7th month, they will review results of the TIDieR survey concerning intervention fidelity (this will be completed by one of the Team Leads in advance of the session) and participate in a focus group discussion, with questions guided by the 2022 NPT framework to discuss the clinic's implementation of I2 using their assigned approach.

Analysis Plan CRC screening outcomes will be monitored for all enrolled patients, and will be extracted from data routinely collected in each participating clinic's electronic medical record. Cleaning and management routines (e.g., logical checks for continuous variables, compliance with skip patterns, missing data codes) will be conducted using SAS v9.4.132, paying attention to the range and distribution of the data. Investigators will examine that distribution for all baseline quantitative measures, cos mparing the clinics assigned to NPT-PLA vs 'usual QI' clinics. The unit of analysis will be individual patients within clinics. Investigators will exclude screening outcomes for patients who participate in the 'implementation teams', since participation on the i-team may bias the patient towards completion of I2 and CRC screening, differently than other clinic patients. Investigator will calculate unadjusted risk ratios and use Chi-squared test (likelihood ratio method) to compare the main outcomes for patients in each treatment arm. They will use means or median tests of equality to assess inequality in age, gender, employment, insurance coverage between NPT-PLA vs usual QI clinics, to determine the effectiveness of randomization procedures to balance these patient-level factors between treatment arms. Demographic data e.g. age and sex will also be extracted from participating clinic EMRs to include in adjusted analytic models of the main outcome responses if, at baseline, there are any differences between treatment group demographics. A priori, investigators will include patient's preferred language.Other variables will be selected for inclusion in the models (if they vary between groups at baseline) by backward elimination procedure using the Bayesian information criterion (BIC). Potential multicollinearity will be examined by variance inflation factor (VIF). Investigators will use linear mixed models using a logistic model (primary screening outcome completed vs not), including a random effects term to account for patients' clinic of origin. Another sensitivity analysis with interactions between included variables and treatment group (NPT-PLA vs Usual QI control) will be examined and used to stratify results if significant. Investigators will report the results of this test for preferred language. They will repeat this analysis for the secondary aim outcome (completion of the I2 tool), as described above; however for this outcome they will use an ordinal logistic model.

For aim 2 outcomes, investigators will use both quantitative and qualitative data. They will follow a similar approach to that described for Aim 1 quantitative analyses. They will analyze pre-post changes in NOMAD construct scores, and compare 6-month NOMAD scores between treatment groups. They will use linear mixed models, analogously to the approach used for Aim 1 outcomes, but (because NOMAD construct scores are quantitative) they will use a Gaussian model. If these scores will not be normally or homogenously distributed between groups, they will use appropriate data transformations so as to enable use of use parametric modeling.

DARTNet staff responsible for qualitative coding will review monthly summaries of clinic "checkin calls" (for which investigators will collect field notes) and graphical material from NPT-PLA clinic PLA sessions. Research staff (PI LeMaster, Co-I MacFarlane and DARTNet staff) are experienced in qualitative analysis, and will examine the qualitative data generated during the study (focus group transcripts, meeting and field notes), as well as PLA and other clinic team meeting notes to identify emerging qualitative themes and how they vary across clinical contexts. Investigators will conduct a deductive framework analysis, structured according to the NPT (2022) construct and using a project specific set of validated coding rules. They will use the newly available empirical coding manual for NPT that includes 12 primary and 16 secondary constructs which are organized into a "Context-Mechanism-Outcome (CMO) structure. These identify, characterize, and explain the course of implementation processes through which strategic intentions are translated into behaviors, and how enactment of those behaviors lead to different outcomes and maintenance of CRC screening practices. This analysis will provide insight into differences in implementation pathways experienced in each treatment group (NPT-PLA vs control). Thus investigators are using an extension of the original NPT model to evaluate the implementation process in each clinic.

The CMO constructs and their cross-walk to NPT constructs are as follows:

* Contexts are events in systems unfolding over time within and between settings in which implementation work is done (primary NPT constructs: strategic intentions, adaptive execution, negotiating capability, reframing organizational logic).
* Mechanisms motivate and shape the work that people do when they participate in implementation processes (primary NPT constructs: coherence-building, cognitive participation, collective action, reflexive monitoring).
* Outcomes are the effects of implementation work in context-that make visible how things change as implementation processes proceed (primary NPT constructs: intervention performance, normative restructuring, relational restructuring, sustainment).

Investigators will identify which of these constructs was dominant across clinics in each arm and during clinic participation; how these were expressed in each and across clinic contexts; and (prior to report completion/results dissemination) discuss these themes with participating implementation team members, to check that their perspectives are taken into account in the analysis.

During the analysis of all qualitative data, investigators will pay active attention to any data that fall outside the NPT constructs to appraise its relevance for understanding the implementation processes. DARTNet staff not involved in the design of the study will undertake the initial coding and refer unclear coding issues to Dr. MacFarlane (who is highly expert in qualitative analysis). After initial coding is completed, these staff will meet with Dr. MacFarlane and the study AnalysisTeam monthly during year 5 of the study to discuss qualitative themes emerging from these data.

Sample size: Investigators base their primary power analysis on the Aim 1 outcome "CRC screening completed", since this is the final endpoint of the implementation of the I2 tool; and "CRC orders completed" must precede "CRC screening completed". Investigators are primarily interested in increases in screening uptake in each study arm. Assuming that the effect size of the intervention is at least that of our 2021-22 pilot study comparing NPT-PLA to usual QI in 4 clinics (2 participated in each arm) in which the proportion overall who completed CRC screening in the NPT-PLA arm=50%, and 37% in usual QI control clinics, Mantel-Haenzsel odds ratio adjusting for language = 1.72 (95% C.I. 1.08 - 2.75), two-sided p=0.02), if investigators recruit 10 NPT-PLA and 10 usual QI control clinics in a cluster randomized trial, and if clinics will each enroll at least 100 patients within 6 months of starting participation, with intra-class correlation coefficient=0.02, the study will have at least 82% power, when using a two-sided test at the 0.05 significance level, to detect a significant difference between arms in the proportion of patients for whom CRC screening is completed .

ELIGIBILITY:
Inclusion Criteria:

Clinics participating in the DARTNet Institute /AAFP-affiliated NRN clinic serving communities in which at least 25% of the population prefers Spanish-language.

Clinic implementation teams Patients participating in implementation teams for whom Spanish is their preferred language, who are bilingual in English and Spanish, Clinics Staff will be included who have any contact regarding CRC screening with patients eligible for screening.

Patients whose CRC screening outcomes will be monitored:

adults 45 to 75 years of age who are due for CRC screening, i.e. who have not received a high-sensitivity fecal occult blood test or a fecal immunochemical test within the past year, fecal DNA testing within 3 years, sigmoidoscopy or barium enema within 5 years, or colonoscopy within 10 years; and who receive primary care at least annually from the site.

Exclusion Criteria:

* patients ineligible for routine screening based on a personal or close family history of colorectal cancer or who have increased genetic risk of colon cancer.
* cognitive or decisional incapacity will be excluded from the implementation teams, after completion of a brief, validate screening tool, the Mini-Cog Exam.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Completion of CRC screening orders | continuously monitored for 6 months after the patient is invited to complete the I2 tool during each clinic's participation month (0-12)
  Extracted from patient participant electronic medical records by DARTNet staff, this will be an indicator variable (0= not completed, 1= completed) indicating if the event occurred within 6 months of the date that the patient was first presented the I2 tool
Aim 1: Completion of recommended CRC screening | Continuously monitored for 6 months after the patient is invited to complete the I2 tool during each clinic's participation month (0-12)
  Extracted from patient participant electronic medical records by DARTNet staff, this will be an indicator variable (0= not completed, 1= completed) indicating if the event occurred within 6 months of the date that the patient was first presented the I2 tool
Aim 2: Summative focus group discussion qualitative data | Month 7 after inception in each clinic
  We have chosen focus group discussions to collect qualitative data in which I-team members will synergistically identify and clarify their views about implementation intervention, as would not take place in individual interviews.
  The purpose of the focus group discussions is to (1) review the TIDieR survey responses to clear up any questions about treatment fidelity (2), review the workflow maps they made in the initial session and discuss how workflow has changed; and (3) explore levers and barriers to work flow changes to implement I2. These focus group discussions will focus on levers and barriers to implementing I2 using the approach that each clinic has used (NPT-PLA or usual QI) using the 2022 NPT framework that accounts for context. We will audiorecord and transcribe and deidentify focus group interview data for qualitative thematic analysis.

SECONDARY OUTCOMES:
Aim 1: Completion of the I2 shared-decision making tool | Continuously monitored for 6 months after the patient is invited to complete the I2 tool during each clinic's participation month (0-12).
  Extracted from a DARTNet-hosted Redcap database into which enrolled I2 results will be recorded, data for this study will be an indicator variable (0= not completed, 1=completed, 2= fully completed) indicating if the event occurred within 6 months after the date that the patient was first presented the I2 tool.
Aim 2: NOMAD Survey | Month 0 and 6 after inception in each clinic
  The NOMAD is a validated survey that includes 23 Likert-style statements (range 0-10) indicating agreement to the statement) corresponding to statements regarding each of the 4 mechanism constructs of the Normalization Process Theory implementation framework. Individual members of the implementation teams in clinics in the NPT-PLA arm of the study will respond to NOMAD to assess the capacity of their clinic to implement the I2 tool and carry out the intervention to which their clinic has been randomized.
Aim 2: Qualitative meeting notes | 0-6 months after inception in each clinic
  NPT-PLA intervention and usual QI control groups will provide reports of their implementation meetings. In NPT-PLA groups this will include a report of of NPT-informed PLA sessions. NPT-PLA Team Leads from each clinic will also DARTNet/AAFP NRN study staff in monthly 'checkin' meetings, during which a staff report will be made . Similar 'checkin' meetings will occur between usual QI control clinic Team leads and a separate study staff member. These minutes will be analyzed with TIDieR checklist data to analyze implementation team fidelity to the assigned arm intervention activities.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W LeMaster, MD MPH, Principal Investigator — University of Kansas; Christina Hester, PhD, Principal Investigator — DARTNet Institute; Keith A Greiner, MD MPH, Principal Investigator — University of Kansas
Locations (1):
- DARTNet Institute, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete NCI-approved data management and sharing plan is available from the contact PI upon request. The data and metadata from this project will be archived at the Inter-university Consortium of Political and Social Research (ICPSR). ICPSR is a CoreTrustSeal certified repository providing long-term access to and preservation of data packages. Access and distribution of data in the data repository from individual enrolled patients will conform to de-identified data set regulations i.e., PHI identifiers will not be included, other than CRC screening order, CRC schedule and completion dates (which will be included as days since enrollment i.e. clinic inception), and participant/enrollee age in years.
  Aim 1 analytic quantitative datasets will include aim 1 outcomes, clinic identifier, study arm, demographic participant/enrollee characteristics, Aim 2 NOMAD survey data, qualitative data from implementation interviews and meetings, and related metadata.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: July 1 , 2025, updates posted every 6 months, once complete no end date
Access Criteria: ICPSR is publicly available. Data cleared by ICPSR for public access have minimal reidentification and harm risk, and therefore, and no restrictions on access. Public data users must protect human subjects' confidentiality by agreeing to ICPSR's Terms of Use. When necessary, ICPSR will work with the research team to protect respondent confidentiality by removing, masking, or collapsing variables in the deposited data to produce a public version of the dataset; however, all PHI will be removed from both quantitative and qualitative data prior to IPD sharing in the data repository.